CLINICAL TRIAL: NCT04658082
Title: A Pilot Trial to Evaluate the Precision and Accuracy of the Non-invasive H.G.R Glucometer
Brief Title: A Pilot Trial of the Non-invasive H.G.R Glucometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Amir Tirosh (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Amir Tirosh, Director, Division of Endocrinology, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sheba-19-6335-at-ctil
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non invasive glucose monitor (Other): Single arm. All subjects will have glucose levels measured both by non invasive glucometer and by core lab
  Interventions: Device: H.G.R (GWave) non-invasive glucometer

INTERVENTIONS:
Device: H.G.R (GWave) non-invasive glucometer — Glucose tolerance test

SUMMARY:
A pilot study evaluating the accuracy of a non-invasive glucose monitor (GWave) with venous glucose measured by core laboratory during a glucose tolerance test (GTT) in patients with type 2 diabetes.

The study is conducted on 5 subjects undergoing a 75gr GTT, with blood glucose measured at baseline and at 8 time points up to 180 minutes post glucose ingestion both by GWave non-invasive glucometer and by core lab glucose measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male or female.
3. Age above or equal to 18 years at the time of signing informed consent.
4. Diagnosed with type 2 diabetes mellitus ≥ 180 days before screening.
5. HbA1c of 6.0-8.0% .

Exclusion Criteria:

1. Participants under the age of 18 years
2. pregnant women or patients with normal blood glucose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
difference between core lab and non invasive glucose measurements | 3 HOURS
  difference between core lab and non invasive glucose measurements

CONTACTS AND LOCATIONS:
Overall Officials: Amir Tirosh, MD PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No